CLINICAL TRIAL: NCT00003342
Title: Phase I Trial of Dose-Dense Gemcitabine, Doxorubicin, Then Paclitaxel Plus Carboplatin In Patients With Transitional Cell Carcinoma of the Urothelium and Impaired Renal Function
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Bladder or Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-114; MSKCC-97114; NCI-G98-1438
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; metastatic transitional cell cancer of the renal pelvis and ureter; localized transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Filgrastim; Carboplatin; Doxorubicin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: doxorubicin hydrochloride
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of giving gemcitabine, doxorubicin, and paclitaxel together with carboplatin in treating patients with advanced bladder or kidney cancer and impaired kidney function.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of dose-dense carboplatin plus paclitaxel on a weekly schedule given in sequence after gemcitabine and doxorubicin in patients with renal impairment and metastatic or locally advanced transitional cell carcinoma of the urothelium.
* Observe the outcome of this sequential systemic chemotherapy in these patients, or following surgical resection as adjuvant therapy in patients in whom poor renal function precludes the use of cisplatin-based chemotherapy.

OUTLINE: This is a dose escalation study of carboplatin.

Patients receive gemcitabine IV over 10 minutes and doxorubicin IV over 15 minutes for 5 doses on weeks 1, 3, 5, 7, and 9. Filgrastim (G-CSF) is given subcutaneously on days 3 through 10 of each 2-week course. On week 11, patients receive paclitaxel and carboplatin IV over 1 hour weekly for 12 weeks.

Each cohort of 3 patients is entered on sequentially increasing doses of carboplatin. If any patient experiences dose limiting toxicity (DLT), then 6 patients are entered at that dose level. If 3 patients experience DLT at any dose level, the maximum tolerated dose has been surpassed and a total of 6 patients are treated at the previous level.

Patients are evaluated at week 16 and at end of study.

PROJECTED ACCRUAL: There will be 18-30 patients accrued into this study over 9-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced transitional cell urothelial cancer

  * Clinical Stage IV: T any, N1-3, M0; T any, N any, M1; or cT4, Nx, M0 (bladder tumors)
  * Pathological Stage III or IV bladder cancer: T any, N1-3, M0; T3b, N0, M0; T4, N0, M0; and T4, Nx, M0
  * Pathological Stage III or IV urothelial cancer of the renal pelvis or ureter: T any, N1-3, M0; T3, N0, M0; T4, N0, M0; and surgery has been performed within 10 weeks of initiation of therapy
* Impaired renal function (See Renal function tests)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100% OR
* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times normal
* Alkaline phosphatase less than 2 times normal
* SGOT less than 2 times normal

Renal:

* Creatinine greater than 1.5 mg/dL but no greater than 2.5 mg/dL OR
* Creatinine clearance 30-59 mL/min

Cardiovascular:

* Normal cardiac function by history, physical examination, and chest radiograph OR
* If prior cardiac disease, left ventricular ejection fraction must be at least 50% by radionuclide ventriculogram or echocardiogram
* No serious cardiac arrhythmias; including first, second, and third degree heart block
* No New York Heart Association class III or IV heart disease

Other:

* No uncontrolled infection
* No other active cancer, except nonmelanomatous skin cancer and in situ carcinoma of the cervix curatively treated
* Not pregnant
* Effective barrier contraception required for all fertile patients during and for 6 months after therapy (encouraged to continue for 2 years or longer)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the bladder
* At least 4 weeks since any other prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean F. Bajorin, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York